CLINICAL TRIAL: NCT06144463
Title: Study on the Application Value of Fluid Resuscitation Guided by Lung Ultrasound in Neonatal Septic Shock
Brief Title: Lung Ultrasound-guided Fluid Resuscitation in Neonatal Septic Shock
Acronym: LUGFRINSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Guangdong Second Provincial General Hospital (Other)
Responsible Party: Principal Investigator, Dabin Huang, Doctor, Guangdong Second Provincial General Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DHuang
Record Dates: First submitted 2023-11-13; First posted 2023-11-22 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Septic Shock
Keywords: Lung ultrasound; fluid resuscitation; neonatal septic shock
MeSH Terms: conditions — Shock, Septic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): No intervention will be given
- traditional group (Sham Comparator): Non-invasive cardiac output monitoring ( NICOM ) assisted fluid resuscitation.
  Interventions: Diagnostic Test: lung ultrasound-guided fluid resuscitation
- LUGFR group (Experimental): lung ultrasound-guided fluid resuscitation
  Interventions: Diagnostic Test: lung ultrasound-guided fluid resuscitation

INTERVENTIONS:
Diagnostic Test: lung ultrasound-guided fluid resuscitation — For the LUGFR group, therapy was applied based on the same treatment guidelines, and initial lung ultrasonography was performed after enrollment as baseline assessment of lung. The lung ultrasound was conducted using the Doppler ultrasound diagnostic instrument (Philips CX50) at a probe frequency range of 8 to 12 MHz. Lung ultrasonography was conducted using the 12-region method that included the anterior, lateral, and posterior walls on both sides of the lung, which was focused on the condition of A-lines, B-lines (including confluent B-line and compact B-lines), lung consolidation and pleural effusion
  Arms: LUGFR group; traditional group

SUMMARY:
object name: Lung ultrasound-guided fluid resuscitation in neonatal septic shock.

type of study: prospective observational study. goal of study: The effects of severe ultrasound-assisted fluid resuscitation and conventional fluid resuscitation on the prognosis of children with neonatal septic shock were compared to evaluate the application value of the two techniques in fluid resuscitation of neonatal septic shock.

research design: In this study, children with neonatal septic shock diagnosed in the neonatal intensive care unit of the Second People 's Hospital of Guangdong Province from January 1,2022 to December 31,2023 were included in the population. According to the different monitoring methods used in conventional / clinical shock treatment, 30 cases of fluid resuscitation assisted by severe ultrasound, 30 cases of fluid resuscitation assisted by NICOM and 30 cases of conventional fluid resuscitation were collected, a total of 90 cases.

( 1 ) The demographic data, blood examination and microbiological examination data of the two groups at admission were collected.

( 2 ) The fluid volume, blood lactic acid, blood pressure, vasoactive drugs ( such as dopamine and epinephrine / norepinephrine ), mechanical ventilation, renal replacement therapy and antibiotic use were collected before fluid resuscitation.

( 3 ) The cumulative fluid infusion volume during fluid resuscitation ( 6 hours ), and the use of vasoactive drugs and mechanical ventilation for 6 hours were collected.

( 4 ) NICU hospitalization time, cumulative hospitalization time and mortality were collected.

Data collection :

( 1 ) The demographic data, blood examination and microbiological examination data of the three groups at admission were collected.

( 2 ) The fluid volume, blood lactic acid, blood pressure, vasoactive drugs ( such as dopamine and adrenaline / norepinephrine ), mechanical ventilation, renal replacement therapy and antibiotic use before fluid resuscitation were collected.

( 3 ) The cumulative fluid infusion volume during fluid resuscitation ( 6 hours ), and the use of vasoactive drugs and mechanical ventilation for 6 hours were collected.

( 4 ) NICU hospitalization time, cumulative hospitalization time and mortality were collected.

DETAILED DESCRIPTION:
Efficacy evaluation: The main efficacy criteria: NICU hospitalization time and cumulative hospitalization time, mortality. Secondary efficacy criteria: cumulative fluid volume during fluid resuscitation (6 hours), and use of vasoactive drugs and mechanical ventilation for 6 hours.

ELIGIBILITY:
Inclusion Criteria:

1. Born less than 28 days on admission ;
2. In line with the diagnostic criteria for neonatal septic shock in the ' 2020 International Guidelines for Saving Sepsis Campaign : Management of Sepsis-related Organ Dysfunction in Children ' ;
3. For children diagnosed with septic shock, fluid resuscitation should be performed according to the routine diagnosis and treatment.
4. The legal guardian has signed the informed consent.

Exclusion Criteria:

1. combined with neurogenic shock, trauma and hemorrhagic shock ;
2. symptomatic patent ductus arteriosus ;
3. combined with congenital heart disease ;
4. give up treatment or death within 24 hours of admission ;
5. The legal guardian refused to participate in the study ;
6. Key information and information missing.

Ages: 1 Day to 28 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
hospitalization time | Within 2 weeks
  Primary indicator
mortality | Within 2 weeks
  Primary indicator

SECONDARY OUTCOMES:
Cumulative fluid volume | Within 2 weeks
  Secondary Outcome
Use of vasoactive drugs | Within 2 weeks
  Secondary Outcome
Use of mechanical auxiliary gas | Within 2 weeks
  Secondary Outcome

CONTACTS AND LOCATIONS:
Overall Officials: Zhenyu Liang, Master, Study Director — Department of Pediatrics, Guangdong Second Provincial General Hospital, Guangzhou, China
Locations (1):
- Guangdong Second Provincial General Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Singh Y, Tissot C, Fraga MV, Yousef N, Cortes RG, Lopez J, Sanchez-de-Toledo J, Brierley J, Colunga JM, Raffaj D, Da Cruz E, Durand P, Kenderessy P, Lang HJ, Nishisaki A, Kneyber MC, Tissieres P, Conlon TW, De Luca D. International evidence-based guidelines on Point of Care Ultrasound (POCUS) for critically ill neonates and children issued by the POCUS Working Group of the European Society of Paediatric and Neonatal Intensive Care (ESPNIC). Crit Care. 2020 Feb 24;24(1):65. doi: 10.1186/s13054-020-2787-9. PMID 32093763
- [Derived] Huang D, You C, Mai X, Li L, Meng Q, Liang Z. Lung ultrasound-guided fluid resuscitation in neonatal septic shock: A randomized controlled trial. Eur J Pediatr. 2024 Mar;183(3):1255-1263. doi: 10.1007/s00431-023-05371-9. Epub 2023 Dec 14. PMID 38095714

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-11-29): https://cdn.clinicaltrials.gov/large-docs/63/NCT06144463/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-29): https://cdn.clinicaltrials.gov/large-docs/63/NCT06144463/ICF_001.pdf